CLINICAL TRIAL: NCT02916849
Title: A Feasibility Study of an Intervention Using a Mobile Application to Promote Strength and Balance and Reduce Risk of Falls in Older People
Brief Title: A Feasibility Study of a Mobile Application Intervention to Promote Strength and Balance Exercises in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: The Swedish Research Council (Other Government); Forte (Industry); Glasgow Caledonian University (Other)
Responsible Party: Principal Investigator, Marlene Sandlund, Assistant Professor, Umeå University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SafeStep
Record Dates: First submitted 2016-09-13; First posted 2016-09-28 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2016-09

CONDITIONS: Accidental Falls
Keywords: Accidental Falls; Prevention & Control; Exercise; Exercise therapy/methods*; Aged; Aged 80 and over; Smartphone; Computers; Computers handheld; Motivation; Postural balance; Health behaviour; mHealth; eHealth
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Safe Step - Health Care Centre (Experimental): Participants will be recruited informed and asked for participation in the study by health care professionals. If included in the study, and choosing the Safe Step exercise program as intervention, participants will be given a green prescription for exercise using the application Safe Step. After an introduction meeting in small groups and pre-assessments the participants will create an individual exercise programme containing ten balance and leg strengthening exercises in the application. During the four month intervention the participants will create weekly exercise plan, keep a digital exercise diary, and receive motivational feed-back within the system. The participants will be recommended to exercise at least three times per week and for at least 30 minutes at a time.
  Interventions: Other: Safe Step
- OEP - Health Care Centre (Active Comparator): Participants will be recruited informed and asked for participation in the study by health care professionals. If included in the study, and choosing the Otago Exercise Program as intervention in the study participants will be given a green prescription for exercise with the Otago Home Exercise Programme-booklet. After an introduction meeting in small groups and pre-assessments the participants will create an individual exercise programme containing ten balance and leg strengthening exercises using the booklet for guidance. During the four month intervention the participants will keep a paper-based exercise diary that will be sent to the researchers on a monthly basis. The participants will be recommended to exercise at least three times per week and for at least 30 minutes at a time.
  Interventions: Other: OEP
- Safe Step - Advertising (Experimental): Participants are recruited through meetings at senior citizens organisations and interviewed by telephone for background data and choice of intervention before inclusion. After an introduction meeting in small groups and pre-assessments the participants will create an individual exercise programme containing ten balance and leg strengthening exercises in the Safe Step application. During the four month intervention the participants will create weekly exercise plan, keep a digital exercise diary, and receive motivational feed-back within the system. The participants will be recommended to exercise at least three times per week and for at least 30 minutes at a time
  Interventions: Other: Safe Step
- Safe Step mentors- Advertising (Experimental): This arm is exactly the same as the Safe Step Advertising group except the participants will be invited to attend group meetings with peer mentors, once a month during the intervention. The peer mentors are older adults earlier involved in the research project . They will act as role models and encourage the participants throughout the four months of exercise.
  Interventions: Other: Safe Step
- OEP - Advertising (Active Comparator): Participants are recruited through meetings at senior citizens organisations and interviewed by telephone for background data and choice of intervention before inclusion. After an introduction meeting in small groups and pre-assessments the participants will create an individual exercise programme containing ten balance and leg strengthening exercises using the Otago booklet for guidance. During the four month intervention the participants will keep a paper-based exercise diary that will be sent to the researchers on a monthly basis. The participants will be recommended to exercise at least three times per week and for at least 30 minutes at a time.
  Interventions: Other: OEP

INTERVENTIONS:
Other: Safe Step — Strength and balance exercise-digital version
  Arms: Safe Step - Advertising; Safe Step - Health Care Centre; Safe Step mentors- Advertising
Other: OEP — Strength and balance exercise -paper version
  Arms: OEP - Advertising; OEP - Health Care Centre

SUMMARY:
This five arm feasibility study aims to promote self-management in strength and balance exercises among community-living older people. The research process, implementation strategies and procedures, acceptability of the exercise programs, perceived benefits of the programs, and the ecological validity, acceptability and ability to detect change of possible outcome measurements will be evaluated before a future randomized controlled trial. A comparison of two exercise programs will be performed; a) Safe Step, a mobile technology based exercise program with motivational strategies, developed by researchers in collaboration with older adults, and b) Otago Exercise Program (OEP), home exercises presented in a booklet. The older participants will be free to select either of the intervention programs and the selection process and outcome will be studied as part of the process evaluation.

The participants in three of the arms (OEP, Safe Step, and Safe Step with mentors) will be recruited through advertisements in local papers and through posters and meetings at senior citizens organisations. In the fourth and fifth arms (OEP and Safe Step) the participants will be recruited from health care centres and their registered professionals with experience of greens prescriptions (Fysisk aktivitet på recept). All five groups, with at least 10 participants in each, will be exercising for four months and will undergo testing at baseline, after two and four months and they will be asked to keep an exercise diary (digital or paper format) during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Independently living
* Able to rise from a high chair
* Able to stand without support
* Experience an impaired balance

Exclusion Criteria:

* Progressive disease that impairs mobility
* Dementia diagnosis
* Intense exercising more than 3 hours / week

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Adherence | after 4 month
  adherence to the program from baseline to four months

SECONDARY OUTCOMES:
Change: Attitudes to Falls-Related Interventions Scale (AFRIS) | baseline, two month and four month
Change: Behavioural Regulation In Exercise Questionnaire (BREQ-2) | baseline, two month and four month
Change: Iconographical Falls Efficacy Scale (Icon-FES) | baseline and four month
  Participants' falls-efficacy in certain situations
Change: Activity Specific Balance Confidence Scale (ABC) | baseline and four month
  Participants' falls-efficacy in certain situations
Change: Late-Life Function and Disability Instrument (LLFDI) | baseline and four month
  a person's ability to do discrete actions or activities, and disability-a person's performance of socially defined life tasks
Change: Short Physical Performance Battery | baseline and four month
  Standing balance, leg muscle strength in chair stand, and gait speed
Change: 30 second chair-stand | baseline and four month
  Leg muscle strength in chair stand
Usability of the programs | Up to four months
  Interviews and observations
Uptake | baseline
  Proportion of invited participants that accepted and started the program.

OTHER OUTCOMES:
Background data | Baseline
  Before the study the participants will fill in a questionnaire with background data containing: self-reported health, medical diagnoses, medication, age, sex, earlier work, computer skill and number of falls previous year.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Sandlund, Ass. Prof., Principal Investigator — Department of Community Medicin and Rehabilitation, 90187 Umeå University, Swewn
Locations (1):
- Caring Science Buildning, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Contact the author. Data will be kept for 10 years after trial finishes.

REFERENCES:
- [Derived] Pettersson B, Janols R, Wiklund M, Lundin-Olsson L, Sandlund M. Older Adults' Experiences of Behavior Change Support in a Digital Fall Prevention Exercise Program: Qualitative Study Framed by the Self-determination Theory. J Med Internet Res. 2021 Jul 30;23(7):e26235. doi: 10.2196/26235. PMID 34328438
- [Derived] Mansson L, Lundin-Olsson L, Skelton DA, Janols R, Lindgren H, Rosendahl E, Sandlund M. Older adults' preferences for, adherence to and experiences of two self-management falls prevention home exercise programmes: a comparison between a digital programme and a paper booklet. BMC Geriatr. 2020 Jun 15;20(1):209. doi: 10.1186/s12877-020-01592-x. PMID 32539711